CLINICAL TRIAL: NCT03243045
Title: Evaluation of Systemic Microvascular Density and Endothelial Function in Patients With Resistant Hypertension After Renal Sympathetic Denervation
Brief Title: Systemic Microvascular Function in Patients With Resistant Hypertension After Renal Sympathetic Denervation
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, MD, PhD, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CAAE-51310815.0.0000.5272
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Arterial Hypertension; Resistant Arterial Hypertension
Keywords: Arterial hypertension; Microcirculation; Sympathetic nervous system
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Renal sympathetic denervation — Transcutaneous renal sympathetic denervation

SUMMARY:
It has been proposed that the modulation of the activity of the sympathetic nervous system, through renal sympathetic denervation, besides reducing blood pressure, would promote an improvement in vascular reactivity and consequent improvement of macro and microcirculation.

The present study aimed to investigate the influence of the renal sympathetic denervation on the skin microvascular function of patients presenting with resistant arterial hypertension.

DETAILED DESCRIPTION:
Arterial hypertension is still a serious public health problem with considerable social and economic impact. Arterial hypertension is the result from a complex interaction between environmental and genetic factors that initiate and perpetuate elevated blood pressure. Studies show that about 10% of patients undergoing treatment have resistant hypertension, defined as high blood pressure refractory to at least three antihypertensive drugs. It is known that the sympathetic nervous system plays a fundamental role in the pathophysiology of hypertension, contributing to metabolic and vascular changes. The sympathetic nervous system has also a major role in the pathophysiology of arterial hypertension. Arterial hypertension has also been associated with functional microcirculatory alterations as well as systemic microvascular endothelial dysfunction in hypertensive patients, confirmed by different microcirculatory flowmetry techniques. In this context, it has been proposed that the modulation of the sympathetic nervous system through renal sympathetic denervation, besides reducing blood pressure, would promote an improvement in vascular reactivity and consequent improvement of macro and microcirculation.

The present study aimed to investigate the influence of the renal sympathetic denervation on the skin microvascular function of patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Resistant arterial hypertension under pharmacological treatment

Exclusion Criteria:

* secondary arterial hypertension
* renal dysfunction
* severe kidney disease
* congestive heart failure

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with a confirmed diagnosis of resistant arterial hypertension who were admitted to the National Institute of Cardiology (NIC) at the Ministry of Health in Rio de Janeiro, Brazil. The NIC is a national reference center for the treatment and research of cardiovascular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Cutaneous microvascular reactivity | Before and one, three, six and twelve months after intervention
  Evaluation of microvascular reactivity using laser speckle contrast imaging
Cutaneous microvascular flow | Before and one, three, six and twelve months after intervention
  Evaluation of the microvascular flow using laser speckle contrast imaging

SECONDARY OUTCOMES:
Cutaneous capillary density | Before and one, three, six and twelve months after intervention
  Evaluation of cutaneous capillary density and reactivity using video-capillaroscopy

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO V TIBIRICA, MD, PhD, Principal Investigator — National Innstitute of Cardiology
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil